CLINICAL TRIAL: NCT07056244
Title: Dexmedetomidine Versus Dexamethasone as Adjuvants to Bupivacaine in Caudal Epidural Block for Pediatrics Undergoing Inguinal Hernia Surgery: A Comparative Prospective Double-Blind Randomized Clinical Trial
Brief Title: Dexmedetomidine Versus Dexamethasone as Adjuvants to Bupivacaine in Caudal Epidural Block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Reham Ragab Younis, Resident-Anesthesia, ICU and pain management department-sohag hospital university, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: soh-Med-25-6-13MS
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: İnguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Dexmedetomidine; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A will receive Bupivacaine + Dexmedetomidine (Active Comparator): Patients will receive Bupivacaine 0.125% at 0.5 ml/kg + Dexmedetomidine 1.5 mcg/kg for post operative analgesia.
  Interventions: Drug: Dexmedetomidine
- group B will receive Bupivacaine + Dexamethasone (Active Comparator): Patients will receive Bupivacaine 0.125% at 0.5 ml/kg + Dexamethasone 0.2 mg/kg for post operative analgesia.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexmedetomidine — as adjuvant to bupivacaine in caudal epidural block for postoperative analgesia
  Arms: group A will receive Bupivacaine + Dexmedetomidine
Drug: Dexamethasone — as adjuvant to bupivacaine in caudal epidural block for postoperative analgesia
  Arms: group B will receive Bupivacaine + Dexamethasone

SUMMARY:
The goal of This prospective, randomized, double-blind comparative study is to compare the efficacy of dexamethasone and dexmedetomidine as adjuvants to bupivacaine 0.125% in caudal epidural block for pediatrics undergoing inguinal hernia surgery, aged 2-6 years.

of Both sex.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-6 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I and II.
* Scheduled for inguinal hernia surgery

Exclusion Criteria:

* Parents or legal guardians refusal.
* Known hypersensitivity to any study drugs.
* Abnormal sacral anatomy
* Local infection at the injection site.
* Neurological disease.
* Coagulopathy.
* Mental retardation.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
duration of postoperative analgesia | "Pain scores will be assessed at 15-minute intervals during the first two hours postoperatively, then at 4, 6, 8,12 and 24 hour"
  FLACC scale (Face, Leg, Activity, Crying, Consolability) total score of 0-10 ,so the duration of analgesia will be defined as the time from caudal injection to the point when FLACC score exceeds 4.

SECONDARY OUTCOMES:
Pain score | "Pain scores will be assessed at 15-minute intervals during the first two hours postoperatively, then at 4, 6, 8,12 and 24 hour"
  Postoperative pain will be evaluated using the FLACC scale (Face, Leg, Activity, Crying, Consolability). Pain scores will be assessed at 15-minute intervals during the first two hours postoperatively, then at 4, 6, 8,12 and 24 hour. The duration of analgesia will be defined as the time from caudal injection to the point when FLACC score exceeds 4, at which time rescue analgesia is needed

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided